CLINICAL TRIAL: NCT02136108
Title: Optimizing Patient Engagement in a Novel Pain Management Initiative (OPEN)
Acronym: OPENtext
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inflexxion, Inc. (Industry)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Lifespan (Other); Rhode Island Hospital (Other); The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Traci Green, Deputy Director, Boston Medical Center Injury Center, Inflexxion, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IHS -1306-02960
Record Dates: First submitted 2014-05-07; First posted 2014-05-12 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Complementary and alternative therapies; Mobile health; Medicaid; Patient navigation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPENtext (Experimental): OPENtext will target cognitive, affective, and behavioral strategies through a single, brief in-person assessment, followed by 12 weeks of theoretically-informed text messages, a core set of information organized in a 'frequently asked questions' structure, interactive peer support, static resources on key patient-identified topics, and a library of peer stories accessible throughout the study period.
  Interventions: Other: OPENtext
- OPENnav (Active Comparator): Peer Navigation is currently offered to some individuals in this Medicaid population but not all. Peer navigators interact with patients by phone/text and at home visits. Efforts focus on drivers of a patient's ED use, and may include providing or identifying patient support, improving health literacy, assisting with transportation vouchers, health education, family support, accessing housing services, and orienting to other community support services.
  Interventions: Other: OPENnav

INTERVENTIONS:
Other: OPENtext — Participants will receive 12 weeks of daily text messages sent from an automated system. The text messages will assist participants in managing their chronic pain.
  Arms: OPENtext
Other: OPENnav — Particpants will be linked with a RIPN PEER Navigator who will assisted them in managing their health care
  Arms: OPENnav

SUMMARY:
The OPEN study has two aims: The first is to identify what helps to keep patients involved with a Medicaid chronic pain management program and to identify features of an ideal text-message-based program for people enrolled in the program. The second aim is to develop the text-message-based program (OPENtext), then find out how useful this intervention is compared to a patient navigator intervention (OPENnav) for increasing patient engagement, improving patient's motivation to manage their chronic pain, and improving patient confidence in self-managing their chronic pain condition.

DETAILED DESCRIPTION:
Chronic pain is a condition that affects the most fundamental aspects of quality of life. Treatment for chronic pain is challenging and usually takes the form of opioid medication therapy. But chronic opioid therapy is also associated with high rates of emergency department use, drug diversion, addiction, and unintentional overdose deaths. The new RI Medicaid Chronic Pain Initiative (CPI) targets patients who are both high emergency department users and experiencing chronic pain. In the CPI, patients can be prescribed an integrated treatment plan of massage, chiropractic, or acupuncture therapies. This is a novel approach to chronic pain care, but retention and patient engagement are low. It is important to understand why involvement in the CPI is low, how to improve the patient experience, and how to support the prescribed CAM therapies.

This study has two aims: The first is to identify what helps to keep patients involved with the CPI program and to identify features of an ideal text-message-based program for people enrolled in the CPI. The second aim is to develop the text-message-based program (OPENtext), then find out how useful this intervention is compared to a patient navigator intervention (OPENnav) for increasing patient engagement, improving patient's motivation to manage their chronic pain, and improving patient confidence in self-managing their chronic pain condition.

Investigators will conduct qualitative interviews with patients, providers, and administrators. Goals of the interviews will be: to understand the patient experience in the CPI, including experiences with the navigation approach currently in place; to identify barriers and facilitators to CPI participation; and to learn how technology-especially cell phone text-messaging-could help support pain care and CPI engagement. These interviews will help develop a text-message-based intervention and provide feedback to existing patient navigator programming. Next, investigators will develop and test the text-message patient support intervention that will contain patient-identified topics and concerns that emerge from the qualitative interviews and topic areas discussed by a stakeholder Advisory Board. Theories of behavior change will be used to help with message development, and patients will take part in helping to test and fine-tune the intervention. Last, investigators will compare the text-message and patient navigation interventions in a randomized controlled study with 200 patients over a six-month period. Investigators will see which approach helps patients increase their involvement in the CPI and better manage their chronic pain. If successful, chronic pain patients across Medicaid programs could benefit from use of the patient navigation or the text-message intervention.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Rhode Island Medicaid Chronic Pain Initiative program

Exclusion Criteria:

* Do not speak English

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Engagement | Once per month for 6 months
  Investigators will capture change in engagement in the CPI program based on utilization of services per month, derived from AMI's administrative records. For the purposes of this study, engagement will be defined as having one or more visits to a CAM provider in a given month.
Readiness to Change | At baseline, 3 months, and 6 months post-randomization
  The Pain Stages of Change Questionnaire (PSOCQ) will be used to measure change in patient's self-reported engagement in the CPI and in the intervention group.
Change in Self-Efficacy | At baseline, 3 months, and 6 months post-randomization
  To measure patient's change in confidence of their ability to self-manage their condition, investigators will use the Chronic Pain Self Efficacy Scale (CPSS).

SECONDARY OUTCOMES:
Pain Severity | At baseline, 3 months, and 6 months post-randomization
  To assess the severity of pain and the impact of pain on daily functions, investigators will use the Brief Pain Inventory short form (BPI), which is commonly used in clinical trials and has documented validity, reliability, and responsiveness to change.
Quality of Life | At baseline, 3 months, and 6 months post-randomization
  Investigators will use the Short Form-12 (SF-12)103, a global measure of patient quality of life with well-established psychometrically sound properties across many disease areas and populations, including chronic pain patients. The SF-12 is responsive to interventions, and is currently being used as the key CPI patient evaluation measure by AMI.
Pain Medication Use | At baseline, 3 months, and 6 months post-randomization
  Schedule II/III opioid medication utilization will derive from the RI Department of Health (HEALTH)'s Prescription Monitoring Program (PMP) database.
Likelihood of Misusing Opioid Medication | At baseline, 3 months, and 6 months post-randomization
  The SOAPP-R and COMM are quick and easy-to-use, designed to help providers evaluate the patients' relative risk for developing problems when placed on long-term opioid therapy (SOAPP-R) or to monitor chronic pain patients on opioid therapy (COMM). As a screening tool, the SOAPP-R and the COMM are recommended by SAMHSA in the treatment of chronic pain in patients with histories of or at risk of substance use disorder.
Safety and Aberrant Pain Medication Use Behaviors | At baseline, 3 months, and 6 month post-randomization
  Investigators will examine patient ED utilization from the health plans' (UH,NH) claims data and prevalence and incidence of aberrant opioid medication use (i.e.,"dr. shopping") from the RI PMP database.
Acceptance & Satisfaction | At 9-month follow up
  Patients will be asked to rate intervention utility and content (relevance, interest) using 5-point Likert scales.

CONTACTS AND LOCATIONS:
Overall Officials: Traci Green, PhD, MSc, Principal Investigator — Inflexxion, Inc., Brown University, and Rhode Island Hospital; Megan Ranney, MD, Study Chair — The Miriam Hospital and Brown University; Elizabeth Donovan, PhD, Study Chair — Independent Consultant
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No